CLINICAL TRIAL: NCT03137693
Title: A Phase II Study of Preoperative Stereotactic Ablative Body Radiotherapy (SABR) for Early-Stage Breast Cancer: Introduction of a Novel Form of Accelerated Partial Breast Radiotherapy
Brief Title: Preoperative Stereotactic Ablative Body Radiotherapy (SABR) for Early-Stage Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no responders/lack of efficacy
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18596
Record Dates: First submitted 2017-04-28; First posted 2017-05-03 (Actual); Results first posted 2020-12-28 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer; Breast Cancer Female; Breast Adenocarcinoma
Keywords: histologically proven; invasive adenocarcinoma of breast; node negative (N0); breast-conserving surgery; negative for Her-2 amplification; estrogen receptor (ER) positive; progesterone receptor (PR) positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy; Radiosurgery; Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Change in Procedure Scheduling (Other): Pre-Surgery SABR: Treatment with Stereotactic Ablative Body Radiation Therapy (SABR) followed by breast-conserving surgery. The usual treatment for patients with early-stage breast cancer who have breast-conserving treatment (BCT) is to receive radiotherapy AFTER surgery, targeting either the whole breast or part of the breast.
  Interventions: Other: Standard of Care Schedule Variation: SABR; Procedure: Breast-conserving Surgery

INTERVENTIONS:
Other: Standard of Care Schedule Variation: SABR — SABR will be delivered over 3 days, prior to surgery.
  Other Names: radiotherapy; Stereotactic Ablative Body Radiation Therapy (SABR)
Procedure: Breast-conserving Surgery — Breast-conserving surgery will be scheduled for 6-8 weeks after SABR and will be conducted by a Moffitt breast surgeon.

SUMMARY:
This study involves a course of radiation to the tumor that is delivered BEFORE surgery. The type of radiation is called stereotactic ablative body radiation therapy (SABR). The purpose of this study is to evaluate the effects, good and/or bad, of pre-operative SABR specifically focusing on its ability to reduce the chances that additional breast surgery will be needed, reducing the amount of breast/heart/lung tissue that is irradiated, and to study the tumor-tissue effects of SABR. The usual treatment for patients with early-stage breast cancer who have breast-conserving treatment (BCT) is to receive radiotherapy AFTER surgery, targeting either the whole breast or part of the breast.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent document prior to conducting any study related assessments or procedures.
* Histologically proven invasive adenocarcinoma of breast.
* Must have marker clip indicating location of target tumor in breast.
* Unifocal tumor less than or equal to 2 cm based on contrast-enhanced prone-breast MRI.
* Must be clinically and radiographically node negative (N0) to participate on this protocol. Clinically suspicious regional nodes by imaging or physical exam require biopsy evaluation to exclude disease involvement.
* Appropriate candidate for breast-conserving surgery based on multi-disciplinary assessment.
* Females age ≥ 50 years.
* Able to tolerate prone body positioning during radiation therapy.
* No prior ipsilateral-breast or thoracic radiotherapy.
* As defined on MRI, target lesion must be at least 10 mm distance from skin (defined as volume encompassing first 3 mm from breast surface).
* Must be estrogen receptor (ER) positive.
* Must be negative for Her-2 amplification. (Either 1+ on semi-quantitative evaluation of immunostain or negative by fluorescent in-situ hybridization).
* No implanted hardware or other material that would prohibit appropriate treatment planning or treatment delivery in the investigator's opinion.
* No history of an invasive malignancy (other than this breast cancer, or non-metastatic basal or squamous skin cancers) in the last 5 years.
* Must not have received nor be planned for neoadjuvant chemotherapy prior to SABR or surgery.
* ECOG performance status less than 2.
* Females of childbearing potential must have a negative urine pregnancy test prior to simulation and within seven days of SABR start.

Exclusion Criteria:

* Have invasive lobular carcinoma.
* Have a Tumor > 2 cm as measured on prone contrast-enhanced breast MRI.
* Have presence of histologically proven lymph node disease.
* Are not a candidate for breast conserving surgery.
* Have had prior ipsilateral-breast or thoracic radiotherapy.
* History of scleroderma or lupus erythematosus with either cutaneous manifestation or requiring active treatment.
* An MRI defined target tumor that is within 10 mm of skin (defined as volume encompassing first 3 mm from skin surface).
* Have amplification of Her-2 (Either 3+ by semi-quantitative immunostain or positive by Fluorescent in-situ hybridization (FISH)).
* Have implanted hardware or other material that would prohibit appropriate treatment planning or treatment delivery in the investigator's opinion.
* History of an invasive malignancy (other than this breast cancer, or non-metastatic basal or squamous skin cancers) in the last 5 years.
* Have received or plan to receive neoadjuvant chemotherapy either before radiotherapy or before surgery.
* A known carrier of BRCA1 or BRCA2 gene mutation.
* Pregnant or unwilling to undergo pregnancy screening.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Montejo, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Liveringhouse CL, Mills MN, Ahmed KA, Washington IR, Lee MC, Khakpour N, Laronga C, Czerniecki B, Soliman H, Weinfurtner RJ, Rosa M, Kim Y, Stringfield O, Abdalah M, Diaz R, Montejo M. Phase 2 Study of Preoperative SABR for Early-Stage Breast Cancer: Introduction of a Novel Form of Accelerated Partial Breast Radiation Therapy. Int J Radiat Oncol Biol Phys. 2023 Jul 1;116(3):611-616. doi: 10.1016/j.ijrobp.2022.12.036. Epub 2023 Feb 15. No abstract available. PMID 36796498
- [Derived] Weinfurtner RJ, Raghunand N, Stringfield O, Abdalah M, Niell BL, Ataya D, Williams A, Mooney B, Rosa M, Lee MC, Khakpour N, Laronga C, Czerniecki B, Diaz R, Ahmed K, Washington I, Montejo M. MRI Response to Pre-operative Stereotactic Ablative Body Radiotherapy (SABR) in Early Stage ER/PR+ HER2- Breast Cancer correlates with Surgical Pathology Tumor Bed Cellularity. Clin Breast Cancer. 2022 Feb;22(2):e214-e223. doi: 10.1016/j.clbc.2021.06.016. Epub 2021 Jul 20. PMID 34384695
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All participants who received Stereotactic Ablative Body Radiotherapy (SABR) prior to breast surgery
Period: Overall Study
Arm/Group | All Participants
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Rate of Pathologic Complete Response (pCR)
Description: Rate of pathologic complete response following pre-operative SABR for early-stage breast carcinoma. pCR: The absence of residual invasive disease in the breast and in the axillary lymph nodes at the completion of the neoadjuvant treatment.
Time Frame: 6 weeks post SABR
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 20
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: 1 year, 11 months
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=20)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Pain (General disorders) | 2 (2)
Infections and Infestations - Other (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT03137693/Prot_SAP_000.pdf